CLINICAL TRIAL: NCT03879772
Title: Dose-Ranging Study of Mometasone Furoate Nasal Spray (SCH 32088) in the Treatment of Children (Ages 6-11) With Seasonal Allergic Rhinitis (Protocol C95-161)
Brief Title: Dose-Ranging Study of Mometasone Furoate (MK-0887/SCH 032088) Nasal Spray in the Treatment of Children (Ages 6-11) With Seasonal Allergic Rhinitis (C95-161)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C95-161; C95-161 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Results first posted 2019-08-12 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- MFNS 25 mcg QD (Experimental): Mometasone furoate nasal spray 12.5 mcg/spray was administered intranasally, one spray per nostril in the morning (upon awakening), daily for 4 weeks. A matching placebo nasal spray was administered intranasally (1 spray per nostril) in the evening. Chlorpheniramine maleate syrup 2 mg/5 mL was to be used for relief of intolerable SAR symptoms.
  Interventions: Drug: Mometasone furoate nasal spray; Drug: Placebo nasal spray; Drug: Chlorpheniramine maleate syrup
- MFNS 100 mcg QD (Experimental): Mometasone furoate nasal spray 50 mcg/spray was administered intranasally, one spray per nostril in the morning (upon awakening), daily for 4 weeks. A matching placebo nasal spray was administered intranasally (1 spray per nostril) in the evening. Chlorpheniramine maleate syrup 2 mg/5 mL was to be used for relief of intolerable SAR symptoms.
  Interventions: Drug: Mometasone furoate nasal spray; Drug: Placebo nasal spray; Drug: Chlorpheniramine maleate syrup
- MFNS 200 mcg QD (Experimental): Mometasone furoate nasal spray 100 mcg/spray was administered intranasally, one spray per nostril in the morning (upon awakening), daily for 4 weeks. A matching placebo nasal spray was administered intranasally (1 spray per nostril) in the evening. Chlorpheniramine maleate syrup 2 mg/5 mL was to be used for relief of intolerable SAR symptoms.
  Interventions: Drug: Mometasone furoate nasal spray; Drug: Placebo nasal spray; Drug: Chlorpheniramine maleate syrup
- BDP 84 mcg BID (Active Comparator): Beclomethasone dipropionate nasal spray 42 mcg/spray was administered intranasally, one spray per nostril in the morning (upon awakening) and in the evening, daily for 4 weeks. Chlorpheniramine maleate syrup 2 mg/5 mL was to be used for relief of intolerable SAR symptoms.
  Interventions: Drug: Beclomethasone dipropionate nasal spray; Drug: Chlorpheniramine maleate syrup
- Placebo (Placebo Comparator): Matching placebo nasal spray was administered intranasally, one spray per nostril in the morning (upon awakening) and in the evening, daily for 4 weeks. Chlorpheniramine maleate syrup 2 mg/5 mL was to be used for relief of intolerable SAR symptoms.
  Interventions: Drug: Placebo nasal spray; Drug: Chlorpheniramine maleate syrup

INTERVENTIONS:
Drug: Mometasone furoate nasal spray — intranasal administration
  Other Names: Nasonex®; MK-0887; SCH 032088
  Arms: MFNS 100 mcg QD; MFNS 200 mcg QD; MFNS 25 mcg QD
Drug: Beclomethasone dipropionate nasal spray — intranasal administration
  Other Names: Vancenase®
  Arms: BDP 84 mcg BID
Drug: Placebo nasal spray — intranasal administration
  Arms: MFNS 100 mcg QD; MFNS 200 mcg QD; MFNS 25 mcg QD; Placebo
Drug: Chlorpheniramine maleate syrup — oral administration
  Other Names: ChlorTrimeton Syrup

SUMMARY:
The purpose of this study was to identify the lowest dosage of mometasone furoate nasal spray (MFNS) that provided adequate efficacy with an acceptable safety profile for children (ages 6-11) with seasonal allergic rhinitis (SAR). The MFNS dose levels of 25, 100, and 200 mcg QD were compared with beclomethasone dipropionate (BDP), as an active control, and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Have at least a one-year history of seasonal allergic rhinitis which previously required treatment for tree and/or grass pollen
* Have a positive skin test response to an appropriate tree and/or grass seasonal allergen within the last year.
* Must be free of any clinically significant disease other than seasonal allergic rhinitis.
* Must be pre-menarcheal.

Exclusion Criteria:

* History of asthma which requires chronic use of inhaled or systemic corticosteroids.
* Current or history of frequent, clinically significant sinusitis or chronic purulent postnasal drip.
* History of rhinitis medicamentosa.
* History of clinically significant nasal candidiasis.
* History of multiple drug allergies or allergy/intolerance to corticosteroids or antihistamines.
* History of upper respiratory tract or sinus infection that required antibiotic therapy within the previous 2 weeks, or viral upper respiratory infection within 7 days prior to Screening.
* History of nasal structural abnormalities, including large nasal polyps and marked septal deviation, that significantly interfere with nasal air flow.
* History of dependence upon nasal, oral or ocular decongestants, or nasal topical antihistamines.
* History of investigational drug use in the last 30 days.
* History of immunotherapy (desensitizing therapy), unless on a stable maintenance schedule for at least one month prior to Screening.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 679 (Actual)
Dates: Start 1996-03-12 (Actual); Primary Completion 1996-07-01 (Actual); Study Completion 1996-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo
Started | 137 | 135 | 133 | 138 | 136
Completed | 133 | 132 | 123 | 130 | 128
Not Completed | 4 | 3 | 10 | 8 | 8
Not completed — Adverse Event | 2 | 2 | 3 | 4 | 3
Not completed — Treatment Failure | 1 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 3 | 1 | 2
Not completed — Did Not Meet Entry Requirements | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo | Total
Number analyzed (Participants) | 137 | 135 | 133 | 138 | 136 | 679
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.8 (1.5) | 8.7 (1.6) | 8.8 (1.6) | 8.7 (1.6) | 8.8 (1.6) | 8.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 54 | 51 | 52 | 260
  Male | 85 | 84 | 79 | 87 | 84 | 419
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 11 | 8 | 8 | 11 | 49
  White | 114 | 111 | 112 | 119 | 113 | 569
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 13 | 11 | 12 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) at Day 8 as Assessed by Investigator
Description: The mean change from baseline at study day 8 was calculated for TNSS as assessed by the investigator. TNSS was a composite of the individual nasal symptom scores of discharge (rhinorrhea), stuffiness, sneezing, and itching. The 4 individual nasal symptom scores were rated by the investigator at the visit as follows: 0=none, 1=mild, 2=moderate, 3=severe. TNSS was the sum of the 4 individual nasal symptom scores (range= 0-12; higher score indicating more frequent/severe nasal symptoms). For each participant, individual scores were totaled and used to calculate the change from Baseline in TNSS at the visit. Participant changes were then used to calculate the mean change for each treatment group at that visit. Change from Baseline = visit score - Baseline score (Day 1 visit). Negative changes indicate a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 8
Population: All randomized participants with a baseline score who completed at least one valid post-baseline visit and had available Day 8 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo
Number analyzed (Participants) | 137 | 135 | 132 | 136 | 134
Scores on a scale
  Baseline | 7.8 (1.7) | 8.1 (1.7) | 7.9 (1.6) | 8.0 (1.7) | 8.0 (1.5)
  Change From Baseline Day 8: number analyzed (Participants) | 133 | 134 | 127 | 134 | 130
  Change From Baseline Day 8 | -2.8 (2.6) | -2.8 (2.6) | -2.8 (2.5) | -2.8 (2.4) | -1.9 (2.2)
Statistical Analysis 1: Comparison: MFNS 25 mcg QD vs MFNS 100 mcg QD; Pairwise comparisons were performed using least square means from two-way analysis of variance (ANOVA); Test type: Superiority; p = 0.95, ANOVA
Statistical Analysis 2: Comparison: MFNS 25 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.78, ANOVA
Statistical Analysis 3: Comparison: MFNS 25 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.98, ANOVA
Statistical Analysis 4: Comparison: MFNS 25 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 100 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.82, ANOVA
Statistical Analysis 6: Comparison: MFNS 100 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.98, ANOVA
Statistical Analysis 7: Comparison: MFNS 100 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.01, ANOVA
Statistical Analysis 8: Comparison: MFNS 200 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.8, ANOVA
Statistical Analysis 9: Comparison: MFNS 200 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.02, ANOVA
Statistical Analysis 10: Comparison: BDP 84 mcg BID vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.01, ANOVA

2. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) on Day 4 as Assessed by Investigator
Description: The mean change from baseline at study day 4 was calculated for TNSS as assessed by the investigator. TNSS was a composite of the individual nasal symptom scores of discharge (rhinorrhea), stuffiness, sneezing, and itching. The 4 individual nasal symptom scores were rated by the investigator at the visit as follows: 0=none, 1=mild, 2=moderate, 3=severe. TNSS was the sum of the 4 individual nasal symptom scores (range= 0-12; higher score indicating more frequent/severe nasal symptoms). For each participant, individual scores were totaled and used to calculate the change from Baseline in TNSS at the visit. Participant changes were then used to calculate the mean change for each treatment group at that visit. Change from Baseline = visit score - Baseline score (Day 1 visit). Negative changes indicate a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 4
Population: All randomized participants with a baseline score who completed at least one valid post-baseline visit and had available Day 4 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo
Number analyzed (Participants) | 137 | 135 | 132 | 136 | 134
Scores on a scale
  Baseline | 7.8 (1.7) | 8.1 (1.7) | 7.9 (1.6) | 8.0 (1.7) | 8.0 (1.5)
  Change From Baseline Day 4: number analyzed (Participants) | 135 | 128 | 128 | 131 | 130
  Change From Baseline Day 4 | -2.2 (2.4) | -2.0 (2.1) | -2.0 (2.5) | -2.4 (2.3) | -1.3 (2.2)
Statistical Analysis 1: Comparison: MFNS 25 mcg QD vs MFNS 100 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.56, ANOVA
Statistical Analysis 2: Comparison: MFNS 25 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.74, ANOVA
Statistical Analysis 3: Comparison: MFNS 25 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.68, ANOVA
Statistical Analysis 4: Comparison: MFNS 25 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 100 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.81, ANOVA
Statistical Analysis 6: Comparison: MFNS 100 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.33, ANOVA
Statistical Analysis 7: Comparison: MFNS 100 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.01, ANOVA
Statistical Analysis 8: Comparison: MFNS 200 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.46, ANOVA
Statistical Analysis 9: Comparison: MFNS 200 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 10: Comparison: BDP 84 mcg BID vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA

3. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) on Day 15 as Assessed by Investigator
Description: The mean change from baseline at study day 15 was calculated for TNSS as assessed by the investigator. TNSS was a composite of the individual nasal symptom scores of discharge (rhinorrhea), stuffiness, sneezing, and itching. The 4 individual nasal symptom scores were rated by the investigator at the visit as follows: 0=none, 1=mild, 2=moderate, 3=severe. TNSS was the sum of the 4 individual nasal symptom scores (range= 0-12; higher score indicating more frequent/severe nasal symptoms). For each participant, individual scores were totaled and used to calculate the change from Baseline in TNSS at the visit. Participant changes were then used to calculate the mean change for each treatment group at that visit. Change from Baseline = visit score - Baseline score (Day 1 visit). Negative changes indicate a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 15
Population: All randomized participants with a baseline score who completed at least one valid post-baseline visit and had available Day 15 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo
Number analyzed (Participants) | 137 | 135 | 132 | 136 | 134
Scores on a scale
  Baseline | 7.8 (1.7) | 8.1 (1.7) | 7.9 (1.6) | 8.0 (1.7) | 8.0 (1.5)
  Change From Baseline Day 15: number analyzed (Participants) | 129 | 133 | 123 | 127 | 128
  Change From Baseline Day 15 | -2.9 (2.7) | -3.0 (2.8) | -3.1 (2.7) | -3.5 (2.8) | -2.4 (2.8)
Statistical Analysis 1: Comparison: MFNS 25 mcg QD vs MFNS 100 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.8, ANOVA
Statistical Analysis 2: Comparison: MFNS 25 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.45, ANOVA
Statistical Analysis 3: Comparison: MFNS 25 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.12, ANOVA
Statistical Analysis 4: Comparison: MFNS 25 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.36, ANOVA
Statistical Analysis 5: Comparison: MFNS 100 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.6, ANOVA
Statistical Analysis 6: Comparison: MFNS 100 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.17, ANOVA
Statistical Analysis 7: Comparison: MFNS 100 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.23, ANOVA
Statistical Analysis 8: Comparison: MFNS 200 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.42, ANOVA
Statistical Analysis 9: Comparison: MFNS 200 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.09, ANOVA
Statistical Analysis 10: Comparison: BDP 84 mcg BID vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.01, ANOVA

4. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) on Day 29 as Assessed by Investigator
Description: The mean change from baseline at study day 29 was calculated for TNSS as assessed by the investigator. TNSS was a composite of the individual nasal symptom scores of discharge (rhinorrhea), stuffiness, sneezing, and itching. The 4 individual nasal symptom scores were rated by the investigator at the visit as follows: 0=none, 1=mild, 2=moderate, 3=severe. TNSS was the sum of the 4 individual nasal symptom scores (range= 0-12; higher score indicating more frequent/severe nasal symptoms). For each participant, individual scores were totaled and used to calculate the change from Baseline in TNSS at the visit. Participant changes were then used to calculate the mean change for each treatment group at that visit. Change from Baseline = visit score - Baseline score (Day 1 visit). Negative changes indicate a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 29
Population: All randomized participants with a baseline score who completed at least one valid post-baseline visit and had available Day 29 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo
Number analyzed (Participants) | 137 | 135 | 132 | 136 | 134
Scores on a scale
  Baseline | 7.8 (1.7) | 8.1 (1.7) | 7.9 (1.6) | 8.0 (1.7) | 8.0 (1.5)
  Change From Baseline Day 29: number analyzed (Participants) | 122 | 127 | 115 | 119 | 120
  Change From Baseline Day 29 | -3.1 (2.9) | -3.7 (2.8) | -3.8 (2.6) | -3.7 (3.0) | -2.5 (2.8)
Statistical Analysis 1: Comparison: MFNS 25 mcg QD vs MFNS 100 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.03, ANOVA
Statistical Analysis 2: Comparison: MFNS 25 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.04, ANOVA
Statistical Analysis 3: Comparison: MFNS 25 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.08, ANOVA
Statistical Analysis 4: Comparison: MFNS 25 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.49, ANOVA
Statistical Analysis 5: Comparison: MFNS 100 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.93, ANOVA
Statistical Analysis 6: Comparison: MFNS 100 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.75, ANOVA
Statistical Analysis 7: Comparison: MFNS 100 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 8: Comparison: MFNS 200 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.71, ANOVA
Statistical Analysis 9: Comparison: MFNS 200 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 10: Comparison: BDP 84 mcg BID vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.01, ANOVA

5. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) [Average of Morning (AM), Evening (PM) Score] Averaged Over Days 1 to 15 as Assessed by Participant
Description: Mean change from baseline (CFB) averaged over study days 1-15 was calculated for TNSS assessed by participants (with assistance from caregiver). Participants scored 4 symptoms (rhinorrhea, stuffiness, itching, sneezing) in diaries using the scale 0=none, 1=mild, 2=moderate, 3=severe. TNSS was the sum of the 4 individual scores (range=0-12; higher score indicating more frequent/severe nasal symptoms.) CFD=the 15-day average score-baseline score. Scores were recorded twice daily, in the morning (AM) and evening (PM). Average AM/PM scores were first calculated separately, then averaged together to obtain the 15-day average score. If diary entries were missing, an average AM or PM score was not calculated. If neither average AM nor PM score were calculated, the total 15-day average score was not calculated. Baseline score=Mean of the Baseline AM (day of visit plus 3 preceding days) and the Baseline PM (3 preceding days) scores. Negative change indicated a decrease in symptom severity.
Time Frame: Baseline and Days 1 through 15 (average over 15 days)
Population: All randomized participants with a baseline score who completed at least one valid post-baseline visit and had available diary data.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo
Number analyzed (Participants) | 137 | 134 | 133 | 137 | 134
Scores on a scale
  Baseline | 6.3 (2.3) | 6.9 (2.4) | 6.9 (2.4) | 6.6 (2.4) | 6.8 (2.5)
  Change From Baseline Days 1 to 15 | -1.5 (2.1) | -1.9 (2.0) | -1.8 (2.1) | -1.9 (2.1) | -1.2 (2.0)
Statistical Analysis 1: Comparison: MFNS 25 mcg QD vs MFNS 100 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.16, ANOVA
Statistical Analysis 2: Comparison: MFNS 25 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.22, ANOVA
Statistical Analysis 3: Comparison: MFNS 25 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.14, ANOVA
Statistical Analysis 4: Comparison: MFNS 25 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.14, ANOVA
Statistical Analysis 5: Comparison: MFNS 100 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.85, ANOVA
Statistical Analysis 6: Comparison: MFNS 100 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.96, ANOVA
Statistical Analysis 7: Comparison: MFNS 100 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 8: Comparison: MFNS 200 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.81, ANOVA
Statistical Analysis 9: Comparison: MFNS 200 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 10: Comparison: BDP 84 mcg BID vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA

6. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) [Average of Morning (AM)/Evening (PM) Score] Averaged Over Days 16 to 29 as Assessed by Participant
Description: as for outcome 5
Time Frame: Baseline and Days 16 through 29 (average over 15 days)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo
Number analyzed (Participants) | 137 | 134 | 133 | 137 | 134
Scores on a scale
  Baseline | 6.3 (2.3) | 6.9 (2.4) | 6.9 (2.4) | 6.6 (2.4) | 6.8 (2.5)
  Change From Baseline Days 16 to 29: number analyzed (Participants) | 134 | 131 | 127 | 135 | 130
  Change From Baseline Days 16 to 29 | -2.1 (2.6) | -2.8 (2.8) | -2.7 (2.7) | -2.6 (2.8) | -1.7 (2.7)
Statistical Analysis 1: Comparison: MFNS 25 mcg QD vs MFNS 100 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.05, ANOVA
Statistical Analysis 2: Comparison: MFNS 25 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.07, ANOVA
Statistical Analysis 3: Comparison: MFNS 25 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.11, ANOVA
Statistical Analysis 4: Comparison: MFNS 25 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.31, ANOVA
Statistical Analysis 5: Comparison: MFNS 100 mcg QD vs MFNS 200 mcg QD; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.94, ANOVA
Statistical Analysis 6: Comparison: MFNS 100 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.73, ANOVA
Statistical Analysis 7: Comparison: MFNS 100 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 8: Comparison: MFNS 200 mcg QD vs BDP 84 mcg BID; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p = 0.79, ANOVA
Statistical Analysis 9: Comparison: MFNS 200 mcg QD vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 10: Comparison: BDP 84 mcg BID vs Placebo; Pairwise comparisons were performed using least square means from two-way ANOVA; Test type: Superiority; p < 0.01, ANOVA

ADVERSE EVENTS:
Arm/Group | MFNS 25 mcg QD | MFNS 100 mcg QD | MFNS 200 mcg QD | BDP 84 mcg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/135 | 0/133 | 0/138 | 0/136
Serious Adverse Events (participants affected / at risk) | 1/137 | 0/135 | 1/133 | 0/138 | 0/136
Other Adverse Events (participants affected / at risk) | 62/137 | 62/135 | 58/133 | 59/138 | 64/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MFNS 25 mcg QD (N=137) | MFNS 100 mcg QD (N=135) | MFNS 200 mcg QD (N=133) | BDP 84 mcg BID (N=138) | Placebo (N=136)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MFNS 25 mcg QD (N=137) | MFNS 100 mcg QD (N=135) | MFNS 200 mcg QD (N=133) | BDP 84 mcg BID (N=138) | Placebo (N=136)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (4) | 3 (5) | 8 (8) | 2 (3)
Nausea (Gastrointestinal disorders) | 7 (13) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 7 (7) | 3 (3) | 5 (6) | 4 (4)
Pyrexia (General disorders) | 7 (7) | 8 (8) | 11 (13) | 10 (11) | 11 (11)
Headache (Nervous system disorders) | 25 (44) | 27 (51) | 22 (28) | 36 (69) | 24 (34)
Asthma (Respiratory, thoracic and mediastinal disorders) | 12 (23) | 10 (28) | 10 (15) | 8 (14) | 17 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 7 (11) | 18 (24) | 11 (18) | 10 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 12 (20) | 6 (8) | 6 (10) | 10 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 6 (7) | 11 (14) | 10 (18) | 12 (15)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 4 (4) | 0 (0) | 2 (4) | 7 (8)

LIMITATIONS AND CAVEATS:
Adverse Event (AE) Preferred Terms were converted from WHO-ART dictionary to the MedDRA version 21.1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator agrees not to publish or publicly present any interim results of the Protocol study without the prior written consent of the Sponsor. The Principal Investigator further agrees to provide thirty (30) days prior to submission for publication or presentation to the Sponsor to review copies of abstracts or manuscripts for publication (including texts of oral presentations) which report any results of the Protocol study.